CLINICAL TRIAL: NCT00405483
Title: A Randomized Controlled Trial Utilizing RSA for a Comparison of Minimally Invasive Surgery (MIS) vs. Standard Exposure in Primary Total Hip Arthroplasty With the ProfemurZ Modular Femoral Stem
Brief Title: RSA for a Comparison of MIS vs. Standard Exposure in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAL06-03
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
Keywords: arthroplasty; RSA; micromotion; osteoarthritis; minimally invasive; ProfemurZ
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally invasive exposure (Active Comparator): Surgical technique, minimal incision
  Interventions: Procedure: Minimally Invasive
- Standard exposure (Active Comparator): Standard Incision
  Interventions: Procedure: Standard exposure

INTERVENTIONS:
Procedure: Standard exposure — Minimal invasive vs standard exposure of the joint is the difference between a small incision, smaller equipment for less tissue damage vs large incision (standard is greater than 10cm)and subsequent more tissue damage.
  Other Names: Surgical technique, standard exposure in hip arthroplasty
  Arms: Standard exposure
Procedure: Minimally Invasive — Minimally invasive surgical technique (minimal incision)
  Arms: Minimally invasive exposure

SUMMARY:
The purpose of this study is to determine if MIS for primary hip replacement surgery increases the risk of long term aseptic loosening as predicted by implant micromotion detected by radiostereometric analysis.

DETAILED DESCRIPTION:
Hip replacement is an effective option for treating chronic hip conditions that cause pain and functional impairment(1). Significant improvements in quality of life, as measured by both disease specific and generic quality of life measures, have been well documented (2-4).

Hip replacement implants are a 'ball in cup' design, and consist of two articulating components: a femoral head replacement which can consist of a ball attached to a stem that is inserted into the proximal femur, and an acetabular component, which can be made of different materials that are inserted into a liner of metal that is inserted into the pelvis. These components can be attached to the patient's bone using either polymethylmethacrylate - a polymer more commonly referred to as bone cement - or by roughening the surface of the implant to allow bone ingrowth. Hip replacements can therefore be broadly classified by the fixation technique used: cemented, uncemented, or hybrid, consisting of a cemented femoral component and an uncemented acetabular component. The uncemented design is very commonly used in younger patients because the quality of bone is better in the patient, the implants have demonstrated long term survival, and the cementing step is no longer necessary for achieving long term fixation.

The 10 year survival of current uncemented total hip designs approaches 95% (5). The majority of the 5% that are revised are done so for aseptic ("non-infected") loosening of the components. The functional results of revision total hip surgery are poorer than primary hip replacement surgery (3, 5, 6). There are approximately 20 000 hip replacement performed each year in Canada (CIHI website); this will result in roughly 1000 revisions over the next 10 years - a great expense, both in terms of health care resources and in patients' loss of function. Obviously, efforts directed at decreasing revision rates are clinically and financially worthwhile.

Implant failure due to aseptic loosening is thought to arise from both patient related factors such as age, sex and diagnosis, and from implant related factors such as design and materials used (5). Efforts at reducing aseptic loosening by changing implant design and cement formulation have occasionally resulted in products that perform well in the laboratory but fail miserably in real life, often after being implanted into large numbers of patients(7-10). This has led to a call for careful and controlled introduction of new implant designs using randomized trials and precise radiographic assessment techniques such as radiostereometric analysis (RSA) to look for early signs of loosening and impending failure (7, 9, 11).

Minimally Invasive Surgery (MIS) is a new technology in the optimization of healthcare services. It has been developed to minimize damage to surrounding tissue during arthroplasty. by reducing the size of the incision. The possible benefit is dramatic reductions in length of stay (LOS) for total hip replacement (THR) patients (12). However, MIS development has led to modifications to existing instrumentation, prostheses and technique which may impact long-term survival of the implant (13). There has been little research investigating the effects of these changes on long-term patient outcomes following MIS surgery. The use of RSA will allow for better understanding of the early fixation of the implant and the potential for early failure due to aseptic loosening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are under the age of 65 years
* Subjects have not had hip replacement surgery on the affected hip
* Subjects have decided to undergo a primary total hip replacement of the affected hip

Exclusion Criteria:

* Having a previous hip infection
* Undergoing surgery for arthritis due to a previous injury, rheumatoid arthritis or hip dysplasia (a hip that did not develop completely)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Primary Completion 2014-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to determine if MIS for primary hip replacement surgery increases the risk of long term aseptic loosening as predicted by implant micromotion detected by radiostereometric analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gross, MD FRCSC, Principal Investigator — Dalhousie University & Capital District Health Authority
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada